CLINICAL TRIAL: NCT05453825
Title: A Phase 2, Multicenter, Open-Label Basket Study of Navicixizumab Monotherapy or in Combination With Paclitaxel or Irinotecan in Patients With Select Advanced Solid Tumors
Brief Title: A Study of Navicixizumab Monotherapy or in Combination in Patients With Select Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OncXerna Theraputics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONCX-NAV-G201
Record Dates: First submitted 2022-07-07; First posted 2022-07-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Triple Negative Breast Cancer; Gastric Cancer; Ovarian Cancer
Keywords: navicixizumab
MeSH Terms: conditions — Colorectal Neoplasms; Triple Negative Breast Neoplasms; Stomach Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Combination navicixizumab + paclitaxel (Experimental): Gastric/GEJ and TNBC cancer patients will be assigned to this treatment arm.
  Interventions: Biological: navicixizumab+paclitaxel
- Combination navicixizumab + irinotecan (Experimental): CRC patients will be assigned to this treatment arm.
  Interventions: Biological: navicixizumab+irinotecan
- Navicixizumab monotherapy (Experimental): CRC,TNBC and ovarian cancer patients will be assigned to this treatment arm.
  Interventions: Biological: navicixizumab monotherapy

INTERVENTIONS:
Biological: navicixizumab+paclitaxel — navicixizumab 3 mg/kg Q2W; paclitaxel 80 mg/m2 weekly
  Arms: Combination navicixizumab + paclitaxel
Biological: navicixizumab+irinotecan — navicixizumab 3 mg/kg Q2W; irinotecan 180 mg/m2 Q2W
  Arms: Combination navicixizumab + irinotecan
Biological: navicixizumab monotherapy — navicixizumab 3 mg/kg Q2W
  Arms: Navicixizumab monotherapy

SUMMARY:
This is a study of navicixizumab monotherapy or in combination with paclitaxel or irinotecan in patients with advanced cancer. Patients will be enrolled into one of the following cancer cohorts:

* Cohort A: CRC
* Cohort B: Gastric and GEJ cancer
* Cohort C: TNBC
* Cohort D: Platinum-resistant/refractory epithelial ovarian, primary peritoneal, or fallopian tube cancer (ovarian cancer)

DETAILED DESCRIPTION:
After completing all screening procedures, including the submission of a tissue sample, patients that meet eligibility requirements will be assigned to receive navicixizumab alone or in combination with another anticancer agent. Treatment is assigned based on the patients type of tumor and the cohort that is open at the time of enrollment. Patients will receive treatment in 4 week cycles, attend study visits and have their heart monitored through echocardiograms and daily blood pressure measurements. Patients will also have their tumors monitored regularly through CT scans. Patients receiving benefit may continue on study drug until their tumor progresses, they experience intolerable side effects, their physician decides it is in their best interest to discontinue therapy or they choose to withdrawal from the study. After discontinuing study treatments, all patients will receive regular follow up calls or visits to assess their status and other anticancer treatments they may start.

ELIGIBILITY:
Inclusion Criteria:

1. Patient provides informed consent.
2. Patient is ≥18 years old.
3. Patient has one of the following locally advanced or metastatic, unresectable solid malignancies that is incurable:

   * CRC
   * Gastric or GEJ cancer
   * TNBC
   * Platinum-resistant/refractory epithelial ovarian, primary peritoneal, or fallopian tube cancer
4. Patient has provided an FFPE archive or newly obtained core or excisional biopsy of a tumor lesion.
5. Patient has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
6. Patient has measurable disease, as defined by RECIST v1.1.
7. Patient has adequate organ function.
8. Female patients of childbearing potential must have a negative pregnancy test.
9. Female patients of childbearing potential must agree to follow instructions for highly effective method(s) of contraception while receiving study treatment and for 6 months after the last dose of study drug.
10. Male patients with female sexual partners of childbearing potential must agree to use an acceptable form of contraception while receiving study treatment and for 6 months after the last dose of any study drug.
11. Patient is willing and able to comply with scheduled visits and procedures.
12. Patient must have discontinued other anticancer interventions before Cycle 1 Day 1 per study protocol.

    Cohort A1 and Cohort A2 - CRC only:
13. Patient has definitive pathologically confirmed adenocarcinoma of the colon or rectum.
14. Patient must have received at least 2 and no more than 3 prior lines of standard therapy for metastatic disease.

    Cohort B1 - Gastric/GEJ cancer only:
15. Patient has definitive pathologically confirmed metastatic gastric or GEJ adenocarcinoma that is not amenable to surgery.
16. Patient must have received only 1 prior line of standard therapy for metastatic disease.

    Cohort C1 and Cohort C2 - TNBC only:
17. Patient has definitive pathologically confirmed metastatic or locally advanced TNBC that is not amenable to surgery or radiotherapy with curative intent.
18. Patient must have received at least 2 prior and no more than 4 prior lines of standard therapy for metastatic disease.

    Cohort D1 - Ovarian cancer only:
19. Patient has definitive pathologically confirmed epithelial ovarian, fallopian tube, or primary peritoneal cancer.
20. Patient must be considered platinum-resistant/refractory.
21. Patient must have received at least 2 and no more than 5 prior lines of standard therapy.

Exclusion Criteria:

1. Patient has cardiac conditions as listed in the protocol.
2. Patient has blood pressure (BP) >140/90 mmHg.
3. Patient is pregnant or lactating.
4. Patient has known untreated, active or uncontrolled brain metastases.
5. Patient with leptomeningeal disease.
6. Patient has a known additional malignancy that was progressing or required active treatment within 2 years prior to the first dose of study medication.
7. Patient has a history of bowel obstruction, including sub-occlusive disease, related to the underlying disease or history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess.
8. Patient has an active infection requiring IV systemic therapy.
9. Patient has known hypersensitivity to any components of any study drug or any of its excipients that, in the opinion of the investigator, suggests a high risk for a severe hypersensitivity reaction while on treatment.
10. Patient has a known clinically significant bleeding disorder.
11. Patient is currently using oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes for which the dose has not been stable for >14 days prior to C1D1.
12. Patient had hemoptysis >2.5 mL within 8 weeks prior to C1D1 or serious bleeding from another site within this time frame.
13. Patient had a major surgical procedure, or significant traumatic injury within 28 days prior to C1D1.
14. Patient has an uncontrolled seizure disorder or active neurologic disease.
15. Patient has a cardiac aneurysm.
16. Patient has a known psychiatric disorder, substance abuse disorder, or geographical travel limitations that in the opinion of the investigator would interfere with patient's ability to cooperate with the requirements of the study.
17. Patient has a history or current evidence of any condition, therapy, or laboratory abnormality that may confound the results of the study, interfere with the patient's participation for the full duration of the study, or indicates a condition for which study participation is not in the best interest of the patient, in the opinion of the investigator.

    Cohort A1 and Cohort A2 - CRC only:
18. Patient has known microsatellite instability-high status.

    Cohort A2 - CRC (navicixizumab + irinotecan) only:
19. Patient is on dialysis.
20. Patient has received hepatic intra-arterial chemotherapy.

    Cohort B1 - Gastric/GEJ cancer only:
21. Patient has experienced weight loss >10% over 2 months prior to first dose of study treatment.
22. Patient has definitive pathologically confirmed HER2 positive metastatic gastric or GEJ adenocarcinoma.
23. Patient has pre-existing Grade ≥2 peripheral neuropathy, according to CTCAE v5.0.

    Cohort C2 - TNBC (navicixizumab + paclitaxel) only
24. Patient has pre-existing Grade ≥2 peripheral neuropathy, according to CTCAE v5.0.

    Cohort D1 - Ovarian cancer only:
25. Patient has non-epithelial ovarian carcinoma.
26. Patient has ovarian tumors with low malignant potential (ie, borderline tumors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 12 months
  The proportion of patients with a confirmed best overall response (BOR) of complete response (CR) or PR by Response Evaluation Criteria in Solid Tumors, version 1.1 as determined by investigator tumor response assessments
Progression Free Survival (PFS) | Up to 12 months
  The time from first dose to the date of first documentation of objective disease progression or death (any cause), whichever occurs first, as determined by investigator tumor response assessments

SECONDARY OUTCOMES:
Adverse Events | Up to 12 months
  Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (CTCAE v5.0); clinical laboratory tests; vital sign measurements; electrocardiograms (ECGs); Doppler echocardiograms (ECHOs); physical examinations (PEs)
Overall Survival (OS | Up to 18 months
  Defined as the time from first dose to death
Time to Response (TTR) | Up to 12 months
  Defined as the time from first dose to first documentation of response (CR or PR)
Disease control rate (DCR) | Up to 12 months
  Defined as the proportion of patients with SD or a confirmed BOR of CR or PR
Duration of Response (DOR) | Up to 18months
  Defined as the time from first documentation of response (CR or PR) to documentation of objective disease progression or death due to any cause, whichever occurs first
Xerna™ TME biomarker | Up to 18 months
  Relationship between antitumor activity of navicixizumab therapy and Xerna™ TME Panel biomarker subtypes

OTHER OUTCOMES:
Cancer antigen-125 response | Up to 12 months
  Serum levels of cancer antigen-125 (CA-125) to determine CA-125 response (Cohort D [ovarian cancer] only) and biomarker research through the analysis of tumor and blood samples
Immunogenicity | Up to 6 months
  The presence of anti-navicixizumab antibodies (ie, immunogenicity)
Navicixizumab Pharmacokinetics | Up to 6 months
  Navicixizumab concentrations by time point

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Keck Medicine of USC, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Hematology Oncology Clinic, Baton Rouge, Louisiana
  - New York University - Langone Health - Perlmutter Cancer Center, New York, New York
  - The Zangmeister Cancer Center, Columbus, Ohio
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No